CLINICAL TRIAL: NCT01428193
Title: Effect of Androgen Blockade on Sensitivity of the GnRH Pulse Generator to Suppression by Estradiol and Progesterone in Hyperandrogenic Adolescent Girls (JCM021)
Brief Title: Effects of Androgen Blockade on Sensitivity of the GnRH Pulse Generator to Suppression by Estradiol and Progesterone
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Haven't enrolled participants since 2010
Sponsor: University of Virginia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, John Marshall, Principal investigator Center for Research in Reproduction, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12632; U54HD028934-18 (NIH)
Record Dates: First submitted 2011-08-29; First posted 2011-09-02 (Estimated); Results first posted 2018-06-04 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Polycystic Ovary Syndrome; Hyperandrogenism
Keywords: PCOS; hyperandrogenemia
MeSH Terms: conditions — Polycystic Ovary Syndrome; Hyperandrogenism | interventions — Flutamide; Progesterone; Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Flutamide, estrace, progesterone (Experimental): For flutamide, subjects weighing > 50 kg will receive 250 mg orally twice a day, and subjects weighing < 50 kg will receive 125 mg orally twice a day for approximately 3 weeks.
  Subjects will be given oral estrace, 0.5-1 mg once a day for 7 days following the first overnight study admission.
  Subjects will be given oral progesterone suspension (20 mg/ml, 25-100 mg) three times a day at 0700, 1500, and 2300 hr for seven days following the first overnight study admission.
  Interventions: Drug: Flutamide; Drug: Progesterone; Drug: estrace

INTERVENTIONS:
Drug: Flutamide — Subjects weighing > 50 kg will receive 250 mg orally twice a day, and subjects weighing < 50 kg will receive 125 mg orally twice a day.
Drug: Progesterone — oral progesterone suspension (20 mg/ml, 25-100 mg) three times a day at 0700, 1500, and 2300 hr for seven days
Drug: estrace — 0.5-1 mg once a day for seven days
  Other Names: (estradiol)

SUMMARY:
The purpose of this study is to understand the effects of elevated male hormones in adolescent girls and how they effect the development of polycystic ovary syndrome (PCOS). If the investigators understand the effects of elevated male hormones levels in girls, the investigators may be able to better treat girls with elevated male hormone levels and perhaps even learn how to prevent the development of PCOS. Females with elevated levels of male hormones respond differently to estrace (estradiol) and progesterone than females with normal male hormone levels. The investigators will be giving you estrogen and progesterone to see how you respond after the male hormone has been blocked by a medication called flutamide.

DETAILED DESCRIPTION:
Similar to women with PCOS, girls with hyperandrogenemia have an increased frequency of LH pulses when compared to age matched controls. An ongoing study by our group is investigating whether the progesterone insensitivity of the GnRH pulse generator in adult women with PCOS is also seen in adolescent girls with hyperandrogenemia. Analysis of the data to date suggests that the hyperandrogenic adolescent girls have decreased hypothalamic progesterone sensitivity when compared to adolescent controls, with a subgroup (consisting of approximately half of the hyperandrogenic girls) having marked progesterone insensitivity similar to that seen in adult women with PCOS. These data have recently been published.

Given that androgens mediate hypothalamic progesterone insensitivity in adult women with PCOS, we hypothesize that androgens play a similar role in adolescent girls with hyperandrogenemia and that progesterone sensitivity can be restored with the use of the androgen receptor blocker flutamide.

Better understanding the effects of hyperandrogenemia in adolescence and its role in the development of PCOS will hopefully lead to improved prevention and treatment strategies for PCOS. This may prove increasingly important if the current epidemic in childhood obesity results in a growing number of girls with elevated androgen levels.

ELIGIBILITY:
Inclusion Criteria:

* Girls ages 13 to 17
* Tanner IV or V stage of puberty
* Post-menarche
* Hyperandrogenemic (total testosterone > 0.4 ng/mL or free testosterone > 35 pmol/L) with or without hirsutism
* Normal aspartate aminotransferase/alanine aminotransferase (AST/ALT) (AST < 35 U/L, ALT < 55 U/L)
* Hemoglobin > 12 mg/dL or Hematocrit > 36%
* Normal screening labs (with exception of the expected hormonal abnormalities inherent in hyperandrogenemia)
* Sexually active subjects must agree to abstain or use double barrier contraception during the study
* Subjects must agree not to take any other medications during the course of the study without approval by the study investigators

Exclusion Criteria:

* Abnormal screening labs (with the exception of the expected hormonal abnormalities inherent in hyperandrogenemia)
* Elevated AST/ALT (AST > 35 U/L, ALT > 55 U/L)
* Hemoglobin <12 mg/dL or hematocrit < 36%
* Weight < 32 kg
* History of liver disease, peanut allergy, deep venous thrombosis, breast cancer, endometrial cancer, or cervical cancer
* Pregnant or breastfeeding
* On medications known to affect the reproductive axis within 3 months of the study (including oral contraceptive pills, metformin, and spironolactone)
* On medications known or likely to inhibit or induce CYP1A2 or CYP3A4 (please see "Restrictions on use of other drugs or treatments" section below for common examples of such drugs)
* Are currently participating in another study or have been in one in the last 30 days.

Ages: 13 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2006-09 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R. McCartney, MD, Principal Investigator — University of Virginia
Locations (1):
- Center for Research in Reproduction, University of Virginia, Charlottesville, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Flutamide, Estrace, Progesterone: For flutamide, subjects weighing > 50 kg will receive 250 mg orally twice a day, and subjects weighing < 50 kg will receive 125 mg orally twice a day for approximately 3 weeks.
  Subjects will be given oral estrace, 0.5-1 mg once a day for 7 days following the first overnight study admission.
  Subjects will be given oral progesterone suspension (20 mg/ml, 25-100 mg) three times a day at 0700, 1500, and 2300 hr for seven days following the first overnight study admission.
  Flutamide: Subjects weighing > 50 kg will receive 250 mg orally twice a day, and subjects weighing < 50 kg will receive 125 mg orally twice a day.
  Progesterone: oral progesterone suspension (20 mg/ml, 25-100 mg) three times a day at 0700, 1500, and 2300 hr for seven days
  estrace: 0.5-1 mg once a day for seven days
Period: Overall Study
Arm/Group | Flutamide, Estrace, Progesterone
Started | 4
Completed | 2
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Elevated screening liver enzymes | 1

BASELINE CHARACTERISTICS:
Arm/Group | Flutamide, Estrace, Progesterone
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants] — Age, Sex/Gender, Race, Ethnicity
  Participants
    <=18 years | 4
    Between 18 and 65 years | 0
    >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 15.5 [14 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Slope of the Percent Change in Luteinizing Hormone (LH) Pulses as a Function of Day 7 Progesterone Level
Description: The primary outcome variable for the study is the slope of the percent change in LH pulses as a function of day 7 progesterone level.
Time Frame: 3 weeks after flutamide treatment
Population: One subject completed the study but had not taken the study medication so her data is unusable. The second subject completed the study. However, no data were formally analyzed. We were subsequently unable to recruit any additional subjects.
Measure: Number; unit: percentage of slope change
Arm/Group | Flutamide, Estrace, Progesterone
Number analyzed (Participants) | 1
percentage of slope change | -0.55

ADVERSE EVENTS:
Time Frame: Two weeks post study drug intervention, at time of last blood draw.
Arm/Group | Flutamide, Estrace, Progesterone
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Flutamide, Estrace, Progesterone (N=4)
Mood change, sadness (Social circumstances) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-20): https://cdn.clinicaltrials.gov/large-docs/93/NCT01428193/Prot_SAP_000.pdf